CLINICAL TRIAL: NCT03657875
Title: Retrospective Study to Describe Prevalence of Hyperkalemia in Russian Population Based on Large Laboratory Network
Brief Title: Retrospective Study to Describe Prevalence of Hyperkalemia in Russian Population Based on Large Laboratory Network (HEKATE)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00280
Record Dates: First submitted 2018-08-27; First posted 2018-09-05 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Hyperkalemia Elevated Plasma K+ Cardiovascular Disease (CVD)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: None Retained — Data collection will be performed from anonymous available database of Independent Laboratory INVITRO.
  For the proper calculation of prevalence proportions and proper assessment of associations, the following method of the selection of tests results for corresponding statistical analysis will be applied:
  * For the analysis of primary endpoint, first available result (chronologically) will always be selected for potassium
  * For the analysis of all secondary endpoints and associations between potassium levels and levels of sodium (Na), eGFR, urine albumin, HbA1C, and NT-proBNP or BNP, chronologically matching results will be selected for potassium and other corresponding parameter, in this case, first available result (chronologically) will be selected for the parameter of interest (i.e. sodium, creatinine (for eGFR), urine albumin, HbA1C, and NT-proBNP or BNP) and matching result (of the same date or ±1 day) for potassium will be selected
  * If any first available result is unreliable o

SUMMARY:
This is a cross-sectional retrospective study of laboratory records of patients who take electrolytes blood tests containing the data of the serum potassium level. This study is an observational one, and there is no intervention into routine clinical practice either in terms of therapy, or special examinations.

ELIGIBILITY:
Inclusion Criteria:

* Males and females tested in the Russian centres of INVITRO laboratory from 01.01.2015 till 31.12.2016;
* 18 years and older;
* Available electrolytes blood test containing of the serum potassium level of the unique patient fits for interpretation.

Exclusion Criteria:

* Blood test cannot be interpreted due to various reasons.
* Blood samples with sing of hemolysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Russia 18 years and older whose blood samples were analysed in the independent laboratory INVITRO for serum potassium level (K), from 01.01.2015 till 31.12.2016.
  From the main dataset with serum potassium level, subgroups will be selected with available serum sodium (Na), creatinine (for calculation of eGFR with CKD-EPI formula), urine albumin, HbA1C, and NT-proBNP or BNP.
Sampling Method: Probability Sample
Enrollment: 53940 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
the proportion of the individuals with the serum potassium level higher than 5.0, 5.5, and 6.0 mmol/L | One day
  To determine the proportion of the individuals with the serum potassium level higher than 5.0, 5.5, and 6.0 mmol/L based on INVITRO laboratory database during 2015-2016 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Invitro, Moscow, Russia